CLINICAL TRIAL: NCT02842671
Title: The Implementation and Evaluation of the Autism Spectrum Ambassador Program
Brief Title: Autism Spectrum Ambassador Program
Acronym: ASAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Cheryl Tierney, Section Chief, Behavior and Developmental Pediatrics, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00004103
Record Dates: First submitted 2016-07-13; First posted 2016-07-25 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; ambassador
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Assigned Ambassador (Intervention Group) (Experimental): Patients who were consented, completed the accommodations survey, and for whom a medical student was available during the time of the the procedure will serve as our intervention group. The participants will be assigned an Ambassador throughout the procedure and will complete a patient satisfaction survey afterwards. The investigators hope to enroll 25 controls.
  Interventions: Other: Assigned Ambassador
- Control Group (No Intervention): Patients who were consented, completed the accommodations survey, but for whom a medical student was not available during the time of the patient's procedure will serve as our control group. The controls will fill out both an accommodations survey before and a patient satisfaction survey after the procedure. No ambassador will be assigned for the procedure day. The investigators hope to enroll 25 controls.

INTERVENTIONS:
Other: Assigned Ambassador — If assigned to the intervention group, participants will be contacted by the assigned medical student ambassador at least 1 day prior to the procedure. A brief discussion will take place to review the child's history and survey results. The family will be met by the Ambassador at the hospital and stay with the family until the patient is in the post anesthesia recovery unit. The ambassador is expected to make accommodations for the child as determined by the accommodations survey results. The family will be required to allow the Ambassador to stay through check-in and the procedure.
  Arms: Assigned Ambassador (Intervention Group)

SUMMARY:
The investigators are evaluating the implementation and the effectiveness of a medical student staffed support program (ASAP) for children diagnosed with Autism Spectrum Disorder coming into Penn State Hershey Children's Hospital for a medical procedure. The ASAP program involves training and assigning a medical student as an Ambassador to help advocate for the special needs of a child with ASD. This study is designed to compare patient satisfaction of children and families who are assigned an Ambassador to those who are not assigned an Ambassador during the procedure. The secondary objectives are to measure overall medical student satisfaction with the program, medical student career interests before and after participation, and medical student comfort level interacting with children with ASD before and after participation.

DETAILED DESCRIPTION:
The Autism Spectrum Ambassador Program (ASAP) is a medical student staffed program designed to improve the experience for children with Autism Spectrum Disorder coming into the Children's Hospital for a day procedure involving anesthesia. This program will pair an interested and trained medical student with a family whose child is scheduled for an outpatient procedure and who is identified as possibly needing special accommodations to improve cooperation and procedure tolerance.

Patients will be identified using the Anesthesia clinic's schedule via PowerChart, consented at the pre-operative anesthesia clinic visit, and enrolled in our program by study personnel. Once enrolled, families will be asked to complete a confidential survey that will identify areas that can be accommodated on the procedure day. Students will gain access to these survey results, contact the family at least 1 day prior to the procedure. A brief discussion will take place to review the child's history and survey results. The student will then create a written, personalized Accommodation Plan to be distributed to personnel and the family. The student will meet the family at the hospital and accompany the family check in until the patient is in the post anesthesia recovery unit.

Students will be trained to chart a child's Accommodation Plan for each member of the treatment team which will be distributed by the student with ample time before the procedure. This accommodation plan will alert each treatment team member including surgical nursing, anesthesia, registration, and to the extent possible surgeons, to what accommodations will be needed to improve the experience of the child. Students will be trained to assist with accommodations by communicating on the family's behalf to hospital personnel to include surgical nursing, anesthesia, registration, and to the extent possible surgeons, among others.

To the extent possible, the investigators hope that having a student advocate, educate staff on the procedure day, and implement changes as needed will improve patient satisfaction with the experience and improve the ease with which a procedure can be carried out for a child with ASD. Students will also be queried as to the experience and survey data will be used to improve the program over time.

Training will be completed so that all members of the treatment team will be aware of the program and aware of the possible accommodations. Treatment team members will be provided additional training to enhance the success of the ASAP program and all treatment team members will be encouraged to work together for the best possible outcome for all patients. Treatment team services include: surgical nursing, anesthesia, registration, and to the extent possible the surgeons involved in the care of these children.

ELIGIBILITY:
Inclusion Criteria:

1. Study participants will be children 30 months to 17 years 2. Study participants will be boys and girls 3. Study participants will have a diagnosis of Autism Spectrum Disorder 4. Study participants will be presenting through the pediatric anesthesia clinic in preparation for a surgical or nonsurgical procedure at the Children's Hospital 5. Study participants must be English Speaking

1. Ambassadors must be enrolled as first, second, third, or fourth year medical students at the Penn State College of Medicine
2. Ambassadors must complete training successfully

Exclusion Criteria:

1. Children under 30 months or older than 17 years
2. Children who do not have a diagnosis of Autism Spectrum Disorder
3. Children who are not having surgery at the Children's Hospital
4. Children who are having a procedure but are not being seen for a pre-anesthesia visit
5. Children who cannot understand and communicate in English

1. Individuals who are not a medical student at the Penn State College of Medicine 2. Medical students who do not complete the training course 3. Medical students who are not deemed appropriate the ASAP Ambassador role as per the discretion of study personnel.

Ages: 30 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction Survey (questionnaire) | 1 year
  Improved patient satisfaction and fewer behavioral complications during the procedure day; data collected using REDCap

SECONDARY OUTCOMES:
Medical Student Satisfaction Survey (questionnaire) | 1 year
  Overall medical student satisfaction with the ambassador program; data collected using REDCap
Medical Student Career Interest (questionnaire) | 1 year
  Medical student career interests before and after participation in this program; data collected using REDCap
Medical Student Comfort Level (questionnaire) | 1 year
  Medical student comfort level interacting with autistic children before and after participation in this program; data collected using REDCap

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Tierney, M.D., Principal Investigator — Developmental Pediatrics
Locations (1):
- Penn State Hershey Children's Hospital, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Gimbler Berglund I, Huus K, Enskar K, Faresjo M, Bjorkman B. Perioperative and Anesthesia Guidelines for Children with Autism: A Nationwide Survey from Sweden. J Dev Behav Pediatr. 2016 Jul-Aug;37(6):457-64. doi: 10.1097/DBP.0000000000000289. PMID 27011004
- [Background] Nayfack AM, Huffman LC, Feldman HM, Chan J, Saynina O, Wise PH. Hospitalizations of children with autism increased from 1999 to 2009. J Autism Dev Disord. 2014 May;44(5):1087-94. doi: 10.1007/s10803-013-1965-x. PMID 24122446
- [Background] Broder-Fingert S, Shui A, Ferrone C, Iannuzzi D, Cheng ER, Giauque A, Connors S, McDougle CJ, Donelan K, Neumeyer A, Kuhlthau K. A Pilot Study of Autism-Specific Care Plans During Hospital Admission. Pediatrics. 2016 Feb;137 Suppl 2:S196-204. doi: 10.1542/peds.2015-2851R. PMID 26908475
- Available data/document: Study Protocol — http://irb.psu.edu
- Available data/document: Informed Consent Form — http://irb.psu.edu — for participants
- Available data/document: Accommodation Survey — http://irb.psu.edu
- Available data/document: Patient Satisfaction Survey — http://irb.psu.edu
- Available data/document: Medical Student Survey — http://irb.psu.edu
- Available data/document: Summary Explanation of Research — http://irb.psu.edu — for medical students